CLINICAL TRIAL: NCT03709485
Title: Analysis of Gut Microbiome in Prostate Cancer Patients
Brief Title: Evaluation of Gut Microbiome in Patients With Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0094-17CTIL
Record Dates: First submitted 2018-10-07; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: microbiome; prostate cancer; sequencing
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prostate biopsy patients (Experimental): a cohort o consecutive patients referred to prostate biopsies. In all patients, a rectal swab will be taken prior to biopsy and antimicrobial treatment. The swab will be cultured and analyzed in the lab for characterization of the microbiome.
  Interventions: Other: rectal swab for microbial culture.

INTERVENTIONS:
Other: rectal swab for microbial culture. — Rectal swab and culture.

SUMMARY:
The research will focus on the possible connection between prostate cancer, and various species of bacteria in the large intestine. In consecutive patients, referred to prostate biopsies, rectal swabs will be taken before the biopsies and before antibiotic treatment. The gut flora will be examined and characterized by a microbiome analysis tool. Negative patients will serve as internal control. The investigators will look for association between prostate cancer of various grades and the presence of specific enteropathogens in the rectal flora of the participants.

DETAILED DESCRIPTION:
Prostate cancer is the no. 1 cancer among men. Risk factors include Afro-American origin, prostate cancer in a first degree relatives and the presence of BRCA2 genetic mutations. No specific association has been described yet between prostate cancer and specific gut bacteria.

The GI tract is the home of billions of bacteria. The microbiome functions as a separate organ and contains 10 times the amount of genes compared to the human genome. The microbiome has crucial impact on the human metabolism, inflammatory processes and filtration of GI content. All of these effects may contribute to the exposure of the human body to various carcinogens and inflammatory factors, leading eventually to the development of cancer in remote organs.

The purpose of this research is to try and identify specific species that might be related to the development of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* age above 45
* referred for prostate biopsy

Exclusion Criteria:

* age below 45
* antimicrobial therapy in the 7 days prior to biopsy
* previous prostate or pelvic irradiation
* patients who suffer from inflammatory bowel disease
* systemic chemotherapy for any reason in the 3 months prior to the biopsy.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males
Enrollment: 150 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of gut microbiome | 1 year
  Analysis of rectal swab cultures.
Association of prostate cancer patients and specific microbes. | 1 year
  Relationship between patients with prostate cancer and specific strains of rectal microbes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liss MA, White JR, Goros M, Gelfond J, Leach R, Johnson-Pais T, Lai Z, Rourke E, Basler J, Ankerst D, Shah DP. Metabolic Biosynthesis Pathways Identified from Fecal Microbiome Associated with Prostate Cancer. Eur Urol. 2018 Nov;74(5):575-582. doi: 10.1016/j.eururo.2018.06.033. Epub 2018 Jul 12. PMID 30007819
- [Background] Golombos DM, Ayangbesan A, O'Malley P, Lewicki P, Barlow L, Barbieri CE, Chan C, DuLong C, Abu-Ali G, Huttenhower C, Scherr DS. The Role of Gut Microbiome in the Pathogenesis of Prostate Cancer: A Prospective, Pilot Study. Urology. 2018 Jan;111:122-128. doi: 10.1016/j.urology.2017.08.039. Epub 2017 Sep 6. PMID 28888753
- [Background] Porter CM, Shrestha E, Peiffer LB, Sfanos KS. The microbiome in prostate inflammation and prostate cancer. Prostate Cancer Prostatic Dis. 2018 Sep;21(3):345-354. doi: 10.1038/s41391-018-0041-1. Epub 2018 May 23. PMID 29795140